CLINICAL TRIAL: NCT01742195
Title: Randomized Study Comparing the Oral and Nasal Routes for Linear Endobronchial Ultrasound
Brief Title: Comparison of Patient Comfort With the Nasal and Oral Insertion of the Endobronchial Ultrasound Bronchoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Antoine Delage, MD, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IUCPQ-20871
Record Dates: First submitted 2012-11-28; First posted 2012-12-05 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Satisfaction
Keywords: Endobronchial ultrasound; Bronchoscopy; Patient satisfaction
MeSH Terms: conditions — Personal Satisfaction; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal EBUS insertion (Other): Patients in this arm will undergo a linear endobronchial ultrasound with the bronchoscope inserted through the nose.
  Interventions: Procedure: Nasal EBUS insertion
- Oral EBUS insertion (Other): Patients in this arm will undergo a linear endobronchial ultrasound with the bronchoscope inserted through the mouth.
  Interventions: Procedure: Oral EBUS insertion

INTERVENTIONS:
Procedure: Oral EBUS insertion
  Arms: Oral EBUS insertion
Procedure: Nasal EBUS insertion
  Arms: Nasal EBUS insertion

SUMMARY:
The aim of this study is to determine if the insertion of the linear endobronchial ultrasound bronchoscope is more comfortable for patients when done through the nose compared to its insertion through the mouth. Our hypothesis is that nasal insertion is more comfortable.

DETAILED DESCRIPTION:
Linear endobronchial ultrasound (EBUS) now plays a crucial role in the diagnosis, staging, and treatment planning of lung cancer. Most centers perform linear EBUS via the oral route given the larger diameter of the bronchoscope used. However, the feasibility and the diagnostic accuracy of linear EBUS performed through the nose have not been reported. Furthermore, the two routes of insertion have never been compared in terms of patient satisfaction and comfort.

In order to compare the two routes of insertion, consecutive patients referred for a linear endobronchial ultrasound will be recruited. Participants will be randomized to either oral or nasal insertion. All participants will be sedated and will receive local anesthetics in a similar manner. After the procedure, patients will fill a questionnaire regarding their comfort and satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years of age
* patients referred for a first linear endobronchial ultrasound

Exclusion Criteria:

* Patients who previously underwent an EBUS
* Patients intubated with an endotracheal tube
* Patients under the age of 18
* Patients unable to provide informed consent
* Patients currently taking anticoagulants (therapeutic doses of intravenous or subcutaneous heparin, low-molecular weight heparins, direct thrombin inhibitors or other agents)
* Patients taking anti-platelet therapy other than aspirin (clopidogrel, ticagrelor, prasugrel). A period of 7 days off medication is required before participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Patient comfort and satisfaction | Two hours after endobronchial ultrasound
  Measured by a questionnaire using a 10-point Likert scale for both comfort and satisfaction.

SECONDARY OUTCOMES:
Physician's assessment of patient comfort | Immediately after the procedure (within 10 minutes)
  Measured by a questionnaire using a 10-point Likert scale regarding patient comfort and procedural difficulties.
Duration of endobronchial ultrasound procedure | During the procedure
  Measured in minutes.
Total doses of sedation | Immediately after the procedure (within 10 minutes)
  Total doses of each sedative used will be recorded.
Occurence of pneumothorax, bleeding more than 50ml, oxygen desaturation to less than 90%, epistaxis, cardiac arrhythmia | During the procedure and up to two hours after
Proportion of adequate cytology specimens in each group | Days after the procedure (results usually available within 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Beaudoin, MD, Principal Investigator — Laval University; Simon Martel, MD, Principal Investigator — Laval University; Antoine Delage, MD, Principal Investigator — Laval University
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Beaudoin S, Martel S, Pelletier S, Lampron N, Simon M, Laberge F, Delage A. Randomized Trial Comparing Patient Comfort Between the Oral and Nasal Insertion Routes for Linear Endobronchial Ultrasound. J Bronchology Interv Pulmonol. 2016 Jan;23(1):39-45. doi: 10.1097/LBR.0000000000000249. PMID 26705010